CLINICAL TRIAL: NCT04578483
Title: Postoperative Pain Management of Therapeutic Surgery: a Prospective, Observational Cohort Study.
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Kee-Ming Man, Director, Department of Anesthesiology, China Medical University Hsinchu Hospital, China Medical University Hospital
Other Study IDs: CMUH109-REC3-101
Record Dates: First submitted 2020-10-05; First posted 2020-10-08 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Pain
Keywords: Postoperative Pain; Analgesics; Analgesia; Dinalbuphine sebacate; Naldebain; PCA; Extended-release
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 16 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ERDS group: Patients receiving one dose of extended-release dinalbuphine sebacate (ERDS) by ultrasound-guided muscle injection will be invited to participate in this study.
  Interventions: Other: ERDS group

INTERVENTIONS:
Other: ERDS group — After anesthesia, extended-release dinalbuphine sebacate (ERDS) is injected into gluteus maximus with ultrasound guidance.

SUMMARY:
Poor management of post-operative acute pain can contribute to medical complications including pneumonia, deep vein thrombosis, infection and delayed healing, as well as the development of chronic. In contrast, appropriate pain control is capable of reducing the postoperative complications, preventing the development of chronic pain, and improving the quality of life. The workloads of medical staffs and health care cost are subsequently decreased. Recently, a lot of analgesic methods have been developed and used in clinical practice, such as patient-controlled analgesia, ultrasound-guided long-term analgesia and multimodal analgesia. This study is aimed to investigate the effect of dinalbuphine sebacate, a long-acting analgesic, in postoperative pain management. This real world data can serve as a reference toward high health care quality.

DETAILED DESCRIPTION:
This is a prospective, observational, cohort study. Patients undergoing elective surgery will be invited to the study. The written informed consent will be obtained prior to participation. Demographic data, underlying condition, surgical procedures, consumption of anesthetics and analgesics, analgesic methods, postoperative complications, pain intensity and life quality will be collected from medical history and by questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 20 to 80.
2. Needing pain management after elective surgery.
3. American Society of Anesthesiology Physical Class (ASA) between 1 and 3.

Exclusion Criteria:

1. Allergic to anesthetics, opioids, or medicine used during study period.
2. Severe comorbidity, such as cardiopulmonary disease and strock.
3. Abuse or long-term use of opioids.
4. Pregnant or breastfeeding.
5. Judged to be unsuitable subjects by investigator.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having elective surgery in China Medical University Hsinchu Hospital were invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 634 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Postoperative pain intensity (numerical rating scale) | From Day 0 to Day 5
  Numerical rating scale (NRS) is used to assess pain intensity from surgical day (Day 0) to five days after surgery (Day 5). NRS is a 11-point scale which labeled from zero (no pain) to ten (worst pain).

SECONDARY OUTCOMES:
Consumption of anesthetics | From Day 0 to Day 5
  Amounts of medicines used during surgery are all analyzed, especially the ones related to analgesia.
Consumption of analgesics | From Day 0 to Day 5
  Amounts of opioids are converted into morphine equivalents. Amounts of NSAIDs are calculated separately.
Adverse events | From Day 0 to Day 5
  Percentage of the population suffering from postoperative adverse events are analyzed, especially the ones related to analgesics.
EQ-5D-5L score | Within 16 weeks after surgery
  EQ-5D-5L questionnaire is used to assess patients' life quality. Patients are asked to fill in the questionnaire prior to surgery, before discharge and/or three months after surgery.
Patient satisfaction | Within 5 days after surgery
  Before discharge, patients are asked to rate satisfaction toward postoperative pain management on a 5-point scale: very satisfied, satisfied, uncertain, dissatisfied, very dissatisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Kee-Ming Man, MD, MS, Principal Investigator — China Medical University Hsinchu Hospital
Locations (1):
- China Medical University Hsinchu Hospital, Hsinchu, Taiwan